CLINICAL TRIAL: NCT01941212
Title: Effect of Music Therapy Intervention on Pain After Gynecological Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMB 017-13
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Pain
Keywords: Music therapy; pain; gynecological surgeries
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Music therapy and Behavioral therapy (Active Comparator): Music and behavioral therapy
  Interventions: Behavioral: Music therapy
- Music only (Active Comparator): Music therapy without behavioral therapy
  Interventions: Behavioral: Music therapy
- Control (No Intervention): Patients will not listen to music neither will get music therapy

INTERVENTIONS:
Behavioral: Music therapy — Music therapy will be given to patients 24 hours prior and for the first 48 hours after surgery
  Arms: Music only; Music therapy and Behavioral therapy

SUMMARY:
To evaluate the effect of musical therapy before and after gynecological surgeries on pain relief following surgery.

The hypothesis is that musical therapy is effective in pain relief following surgical procedures.

DETAILED DESCRIPTION:
The intention with the study is to focus on the first postoperative phase in a case of pain upon gynecologic abdominal surgery. The literature search revealed studies reporting that participates who had pre-operative session of music intervention for relaxation experienced a greater level of reducing pain levels both pre and post their operation than in the participates in the control group. It is therefore a decision to include one pre operative session of intervention with music therapy in the design.

The study will carry out at the Gynecologic Unit, in Rambam Hospital, Israel.

ELIGIBILITY:
Inclusion Criteria:

* Women are schedule to undergo gynecological surgeries

Exclusion Criteria:

* Neuropathy
* Neurological conditions
* Diabetes

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Pain level following surgery | 48 hours following suegery
  VAS will be used for the evaluation of pain level

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, MD, MS, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel